CLINICAL TRIAL: NCT03313843
Title: Prospective Cross Sectional Study To Assess The Clinical Utility of Optical Coherence Tomography to Measure Axonal Degeneration of the Optic Nerve, in a Cohort of 200 Subjects Meeting the Diagnostics Criteria of Multiple Sclerosis
Brief Title: Study to Assess OCT: RNFL and GCL in MS Patients
Status: Completed | Type: Observational
Sponsor: Tampa Bay Uveitis Center, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: TBUC10022017
Record Dates: First submitted 2017-10-09; First posted 2017-10-18 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis
Keywords: Optical Coherence Tomography
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect preliminary data on retinal nerve fiber layer and ganglion cell layer damage in multiple sclerosis (MS) patients, using optical coherence tomography (OCT). For this study the Zeiss Cirrus OCT Imaging System will be used. The same system will be used consistently for the duration of the study.

DETAILED DESCRIPTION:
Hypothesis: Multiple sclerosis results in axonal degeneration which can be assessed objectively and non-invasively by serial OCT measurements of the RNFL and GCL.

This will be a prospective cross-sectional, non-interventional study; total recruitment will be 200 subjects. Recruitment will be stratified to enroll at least 50 subjects currently taking Lemtrada and 50 subjects with a documented diagnosis of ON. The study will enroll subjects primarily from practices in the Tampa Bay Area and adjacent counties. It is a planned non-interventional study; subjects will be followed by their neurologist and the study ophthalmologist and will receive standard of care. All subjects will have the ophthalmological examination and diagnostic measures, by the Principal Investigator, Dr. Grace Levy-Clarke, at Tampa Bay Uveitis Center.

Study Duration: The study duration will be 24 months, with an interim analysis at 50% recruitment status.

There are two primary aims of this longitudinal observational study:

1. To determine whether atrophy within specific retinal layers over time is associated with clinical neurological progression of MS
2. To determine whether an ON history affects the relationship described in aim # 1

Eye Exam: Subject will have an eye exam, including:

Visual Acuity Testing Color Vision Testing Automated perimetry/Peripheral Vision Testing Completing the National Eye Institute Visual Functioning Questionnaire (NEI/VFQ) Slit Lamp Examination Measurement of Intraocular Pressure (IOP) Dilated Fundus Examination (Ophthalmoscopy) Fundus Photography Optical Coherence Tomography: RNFL and Macular OCT

Neurologic Assessments: Must be performed no more than 60 days prior to screening/assessment Day 0 Ophthalmic Assessments

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Pregnant women will be excluded by self declaration
* Male or female
* A diagnosis of MS, that meets the 2010 Revised McDonald Diagnostic Criteria
* A visual acuity of 20/400 or better in at least one eye

Exclusion Criteria:

* Any ocular disease than prevents assessment of the optic nerve and macula by OCT
* Advance glaucoma with optic nerve damage
* Any optic neuropathy not diagnosed as ON associated with MS
* A diagnosis of Macular Degeneration
* Any previous ocular trauma
* Any medical history of a cerebrovascular accident
* Any planned ocular or systemic elective surgery during study duration
* Any contraindication to a comprehensive dilated ophthalmic examination
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients meeting the diagnostic criteria of multiple sclerosis. Patients will be 18 years or older and pregnant women will be excluded. male and fmale patients will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Retinal Nerve Fiber Layer measurement (RNFL: peri-papillary OCT) | Assessed at Baseline then 6, 12, 18 and 24-month time points
  Optical Coherence Tomography (OCT) will be used to assess change in RNFL of patients with multiple sclerosis

SECONDARY OUTCOMES:
Ganglion Cell Layer measurement (GCL: Macular OCT) | Assessed at Baseline then 6, 12, 18 and 24 - month time points
  Optical Coherence Tomography (OCT) will be used to assess change in GCL of patients with multiple sclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Grace Levy-Clarke, M.D., Principal Investigator — Tampa Bay Uveitis Center, LLC
Locations (2):
- United States (2):
  - Tampa Bay Uveitis Center, New Port Richey, Florida
  - Tampa Bay Uveitis Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No